CLINICAL TRIAL: NCT01065285
Title: Evaluation of Vaccination Against Influenza (Seasonal and H1N1) in Patients Presenting Systemic or Autoimmune Diseases Treated or Not With Steroids, and/or Immunosuppressant, and/or Biotherapy: an Open, Prospective Trial (MAIVAX)
Brief Title: Vaccination Against Influenza in Autoimmune Diseases
Acronym: MAIVAX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P 090901
Record Dates: First submitted 2009-10-21; First posted 2010-02-09 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Autoimmune Diseases
Keywords: Influenza; autoimmune diseases; vaccination; H1N1
MeSH Terms: conditions — Autoimmune Diseases; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Evaluation of vaccines against flu (Experimental): Evaluation of vaccines against flu
  Interventions: Biological: Evaluation of vaccines against flu

INTERVENTIONS:
Biological: Evaluation of vaccines against flu — evaluate efficacy and tolerance
  Other Names: Evaluation of vaccines against flu in auto-imune diseases

SUMMARY:
The project is to evaluate immunogenicity, efficacy and tolerance of vaccination against influenza (seasonal and H1N1) in patients affected with systemic and autoimmune diseases.

DETAILED DESCRIPTION:
This prospective study concentrates on patients with vasculitis, systemic sclerosis, Sjögren's syndrome, systemic lupus erythematosus and other connective tissue diseases.

Patients responding to the inclusion criteria, will receive vaccine against seasonal influenza then, 3 weeks later, vaccine against H1N1 influenza. According to the results of ongoing trials a second injection of H1N1 vaccine has been scheduled 3 weeks later. At each consultation a blood sample will be taken to evaluate immunogenicity of vaccination. Two additional consultations have been scheduled: one month after the last vaccine administration and at 6 month, in order to evaluate the occurrence of late side effects.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients presenting autoimmune and systemic diseases,
* treating or not with steroids, and/or immunosuppressants and/or biotherapies, especially vasculitis, scleroderma, Sjogren's syndrome and systemic lupus (main groups)

Exclusion Criteria:

* Absence of informed consent
* Disease which did not responded to the above criteria
* Active infection at time of vaccination
* HIV infection
* History of Guillain-Barre syndrome
* Allergy to one component of the vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Protection against H1N1 influenza, defined by antibody level of 1/40, measured by hemagglutination, 3 weeks after the first injection and after the second injection | 3 weeks
  Mesure of antibody level of 1/40, measured by hemagglutination, 3 weeks after the first injection and after the second injection

SECONDARY OUTCOMES:
Antibody levels against H1N1 in the different groups of patients, defined according diseases and their treatment (comparison of patients treated by immunosuppressants or not treated) | 3 weeks
  Antibody levels against H1N1 in the different groups of patients, defined according diseases and their treatment
Number of side effects related to vaccination | 3 weeks
Number of local side effects related to vaccination (erythema and/or pain at injection site) | 3 weeks
Number of patients who will develop influenza despite vaccination | 3 weeks
Number of patients who had antibodies against H1N1 before vaccination | 3 weeks
Number of hospitalisations and deaths related to influenza | 3 weeks
Number of flares of the autoimmune diseases that could be related to vaccination | 3 weeks
Determine if the induction of LT-CD4 to J21-28 anti-jams is correlated to the concentrations of antibody anti-vaccines measured in 6 months | 18 months
Determine if the basal concentrations of LT-CD4 anti-jam to J21-J28 are correlated to the concentrations of antibody anti-vaccines measured in 6 months | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Loïc GUILLEVIN, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Cochin, Paris, France

REFERENCES:
- [Result] Kostianovsky A, Charles P, Alves JF, Goulet M, Pagnoux C, Le Guern V, Mouthon L, Krivine A, Villiger P, Launay O, Guillevin L; French Vasculitis Study Group. Immunogenicity and safety of seasonal and 2009 pandemic A/H1N1 influenza vaccines for patients with autoimmune diseases: a prospective, monocentre trial on 199 patients. Clin Exp Rheumatol. 2012 Jan-Feb;30(1 Suppl 70):S83-9. Epub 2012 May 11. PMID 22640652